CLINICAL TRIAL: NCT00712712
Title: Evaluation of the Effectiveness of the Radiofrequency Ablation for Reducing Refractory Pain From Bone Metastases
Brief Title: Morphine After Radiofrequency Ablation of Painful Bone Metastases in Patients With Cancer
Acronym: MEDOR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IB-2007-16; IB-MEDOR (Other: Institute Bergonie); INCA-RECF0498 (Other Grant/Funding Number: INCA); 2007-002686-13 (EudraCT Number)
Record Dates: First submitted 2008-07-09; First posted 2008-07-10 (Estimated); Results first posted 2021-03-26 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2021-03

CONDITIONS: Metastatic Cancer; Pain; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: bone metastases; unspecified adult solid tumor, protocol specific; pain
MeSH Terms: conditions — Neoplasm Metastasis; Pain | interventions — Acetaminophen; Morphine; Radiofrequency Ablation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient who has undergone radiofrequency ablation of bone metastases (Experimental): Patient who has undergone radiofrequency ablation of bone metastases, localized, causing pain refractory to radiotherapy or not accessible to new irradiation, biphosphonates and well-conducted morphine analgesic treatment.
  Interventions: Drug: Acetaminophen; Drug: Morphine Sulfate; Other: Questionnaire administration; Procedure: Quality-of-life assessment; Procedure: Radiofrequency ablation

INTERVENTIONS:
Drug: Acetaminophen — Intravenous administration of paracetamol (4 g / 24h) and patient-controlled analgesia (PCA).
  Other Names: Paracetamol
Drug: Morphine Sulfate — Patient-controlled analgesia (PCA), allowing morphine consumption to be titrated to the patient's needs and thus allowing morphine doses to be adapted to an increase in pain in the patient's post-operative period or a rapid analgesic effect of radiofrequency.
  Other Names: Oral morphine equivalent
Other: Questionnaire administration — Pain notebook will allow the patient to describe the pain specific to the metastasis concerned, containing information on :
  * The intensity of the minimum, average and maximum pain of the last 24 months. hours as well as the intensity of the pain of the moment according to a scale 11-point digital,
  * the background morphine analgesic treatment during the last 24 hours,
  * the morphine analgesic treatment taken during painful attacks,
  * the possible undesirable effects of morphine treatment.
  * the morphinic, non-morphinic and co-antalgic treatment is noted, as well as that the total dose of oral morphine or oral morphine equivalent
Procedure: Quality-of-life assessment — Patients' quality of life will be assessed using the quality of life questionnaire EORTC QLQ-C30 at inclusion in the study and at 8 weeks after radiofrequency. ablation.
Procedure: Radiofrequency ablation — Recent technique of thermal destruction of tumors.
  This technique consists of inserting an electrode needle into the tumour under X-ray or ultrasound guidance or intraoperatively under laparoscopy for example. This needle carries a current or a light wave depending on the characteristics of the generator to which it is connected (radiofrequency, laser).
  Radio frequencies are radiation non-ionising electromagnets. In this context of tissue ablathermia wavelengths ranging from 400kHz to 500kHz.

SUMMARY:
RATIONALE: Morphine may reduce pain in patients who have undergone radiofrequency ablation to remove bone metastases.

PURPOSE: This phase II trial is studying how well morphine works after radiofrequency ablation of painful bone metastases in patients with cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Measure the efficacy of morphine sulfate at 8 weeks after radiofrequency ablation (RFA) of bone metastases.

Secondary

* Assess minimum and average pain and analyze use of morphine sulfate before and after RFA.
* Determine disease progression by CT scan of bone.
* Evaluate the percentage of relief associated with RFA, specifically patient satisfaction, quality of life, anxiety, depression, and physical performance during RFA.
* Assess complications and side effects related to RFA and the evolution of possible side effects associated with morphine sulfate therapy.

OUTLINE: This is a multicenter study.

Patients complete a pain questionnaire over 1 week before undergoing radiofrequency ablation (RFA). Patients also complete questionnaires about pain, physical performance, quality of life (QOL), and anxiety at baseline.

Bone metastases are removed by radiofrequency ablation (RFA). After surgery, patients receive acetaminophen and patient-controlled analgesic (PCA) morphine sulfate. PCA morphine sulfate continues with a dose increase of 50% bolus every 24 hours. Patients with maximum pain less than or equal to that at inclusion receive standard morphine sulfate therapy instead.

Data concerning the total dose of PCA morphine sulfate; minimum, average, and maximum pain intensity; side effects and complications of RFA; and total dose of morphine sulfate (or equivalent) is collected daily.

Pain is assessed at 4 and 8 weeks after RFA. Patients complete follow-up questionnaires about physical performance, QOL, and anxiety at 12 weeks. Patients also undergo a CT scan at 12 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed cancer

  * Primary or unknown origin
* Painful bone metastases despite radiotherapy or symptomatic relapse into previously irradiated area with no possibility of repeating radiotherapy

  * Bone metastases may have been treated with bisphosphonates
  * Osteolytic bone or joint (lytic and condensed) confirmed by CT scan and meeting the following criteria:

    * Lesion size ≤ 5 cm
    * No more than 2 painful bone metastases

      * If 2 lesions are to be treated, distinct anatomical locations can be treated at the same time
    * Metastatic bone lesions of the pelvis, sacrum (in absence of canal involvement), ribs, or long bones allowed
  * Pain located at the tumor or in the area
* Maximum pain in the last 24 hours > 4 points (numerical scale to 11 points)

PATIENT CHARACTERISTICS:

* Life expectancy > 3 months
* Platelet count > 50,000/μL
* Prothrombin < 50%
* Activated cephalin time ≤ 1.5 times normal
* Not pregnant
* Fertile patients must use effective contraception
* No geographical, social, or psychiatric reason that would preclude follow up

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy
* At least 3 weeks since prior chemotherapy or bisphosphonates
* At least 1 week since beginning new painkiller therapy or anticoagulation treatment
* More than 30 days since participation in another drug study
* More than 30 days since prior surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2007-12-24 (Actual); Primary Completion 2016-02-11 (Actual); Study Completion 2016-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Florence Dixmerias, MD, Study Chair — Institut Bergonié
Locations (1):
- Institute Bergonié, Bordeaux, France

REFERENCES:
- See also: National Cancer Institute — http://www.e-cancer.fr/Professionnels-de-sante/Le-registre-des-essais-cliniques/Le-registre-des-essais-cliniques/Etudes-cliniques/MEDOR-Essai-de-phase-2-evaluant-l-efficacite-antalgique-de-l-ablation-par-radiofrequence-de-metastases-osseuses-chez-des-patients-ayant-des-metastases-osseuses-a-l-origine-de-douleurs-refractaires-aux-traitements.-essai-clos-aux-inclusions
- See also: KUSAJILI — https://www.kusajili.fr/fr/Trial/Index/2c4d5bcb-216b-4100-8bc5-d6de01527548

RESULTS

PARTICIPANT FLOW:
Groups:
- Patient Who Has Undergone Radiofrequency Ablation of Bone Metastases Localized Causing Pain: Bone metastases refractory to radiotherapy or not accessible to new irradiation, biphosphonates and well-conducted morphine analgesic treatment.
Period: Overall Study
Arm/Group | Patient Who Has Undergone Radiofrequency Ablation of Bone Metastases Localized Causing Pain
Started | 78
Completed | 55
Not Completed | 23
Not completed — Protocol Violation | 11
Not completed — Radiofrequency not done | 3
Not completed — Death | 8
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Patient Who Has Undergone Radiofrequency Ablation of Bone Metastases
Number analyzed (Participants) | 78
Age, Continuous [Median (Standard Deviation); unit: years] | 66 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 78

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Maximum Pain Level Decreased by ≥ 2 Points at 2 Months After Radiofrequency Ablation (RFA)
Description: Difference in maximum pain scores between inclusion and 2 months after radiofrequency ablation (RFA) according to an 11-point numerical scale
  Rate of patients with a decrease of two or more points in their most intense pain, 2 months after the radiofrequency ablation.
  This rate is calculated for the evaluable population for the principal outcome measure.
  This rate is equal to the ratio of the number of patients with a decrease of two or more points in their maximum pain divided by the size of the evaluable population.
  The response rate considered acceptable is 50%, above this threshold the treatment will be considered potentially effective and may be proposed in phase III.
Time Frame: 2 months after radiofrequency ablation (RFA)
Population: Pre-selected patients meeting the inclusion and exclusion criteria. Excluded patients who died, were lost to follow-up, or dropped out of the study within eight weeks after radiofrequency.
  If 25 patients or more are observed with pain reduction of 2 or more points, then the treatment will be considered potentially effective.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Patient Who Has Undergone Radiofrequency Ablation of Bone Metastases
Number analyzed (Participants) | 55
percentage of participants | 83.6 [73.9 to 93.4]

2. Secondary Outcome: Difference in Maximum Pain Scores Between Inclusion and 2 Months After Radiofrequency Ablation
Description: Difference in maximum pain scores between inclusion and 2 months after radiofrequency ablation (RFA) according to a discrete 11-points numerical scale.
  Increased/decreased pain is considered as a variation of at least one point on the numerical scale.
  If 25 patients or more are observed with pain reduction of 2 or more points, then the treatment will be considered potentially effective.
Time Frame: Inclusion and 2 months after radiofrequency ablation (RFA)
Population: Pre-selected patients meeting the inclusion and exclusion criteria. Excluded patients who died, were lost to follow-up, or dropped out of the study within eight weeks after radiofrequency.
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Who Has Undergone Radiofrequency Ablation of Bone Metastases
Number analyzed (Participants) | 55
Participants
  Increased pain | 4
  Unchanged pain | 2
  Decreased pain | 49

3. Secondary Outcome: Intensity of Pain (Minimum, Average, Maximum)
Description: According to a discrete 11-points numerical scale which ranges from 0 (low pain) to 11 (intense pain), intensity of pain (Minimum, Average, Maximum) has been evaluated at different time point between pre-selection and up to 3 months after radiofrequency.
  Assessment of intensity of pain has been done in this order at:
  * Pre-selection visit: First algology assessment within a week (± 3 days) after the radiology consultation,
  * Inclusion visit: Second algology assessment (One week after the first algology assessment)
  * J-1: one day before radiofrequency
  * J+1: One day after radiofrequency
  * Discharge from hospital
  * 7 days after discharge from hospital
  * 1 month after radiofrequency
  * 2 months after radiofrequency
  * 3 months after radiofrequency
  Here, are presented only data collected at the pre-selection visit.
Time Frame: First algology assessment at pre-selection visit
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Patient Who Has Undergone Radiofrequency Ablation of Bone Metastases
Number analyzed (Participants) | 55
score on a scale
  Minimal pain | 0.5 (1.9)
  Average pain | 5.0 (1.9)
  Maximum pain | 8.0 (1.4)

4. Secondary Outcome: Intensity of Pain (Minimum, Average, Maximum)
Description: According to a discrete 11-points numerical scale which ranges from 0 (low pain) to 11 (intense pain), intensity of pain (Minimum, Average, Maximum) has been evaluated at different time point between pre-selection and up to 3 months after radiofrequency.
  Assessment of intensity of pain has been done in this order at:
  * Pre-selection visit: First algology assessment within a week (± 3 days) after the radiology consultation,
  * Inclusion visit: Second algology assessment (One week after the first algology assessment)
  * J-1: one day before radiofrequency
  * J+1: One day after radiofrequency
  * Discharge from hospital
  * 7 days after discharge from hospital
  * 1 month after radiofrequency
  * 2 months after radiofrequency
  * 3 months after radiofrequency
  Here, are presented only data collected at the inclusion visit.
Time Frame: Second algology assessment at inclusion visit
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Patient Who Has Undergone Radiofrequency Ablation of Bone Metastases
Number analyzed (Participants) | 55
score on a scale
  Minimal pain | 2.0 (2.0)
  Average pain | 5.0 (1.8)
  Maximum pain | 8.0 (1.4)

5. Secondary Outcome: Intensity of Pain (Minimum, Average, Maximum)
Description: According to a discrete 11-points numerical scale which ranges from 0 (low pain) to 11 (intense pain), intensity of pain (Minimum, Average, Maximum) has been evaluated at different time point between pre-selection and up to 3 months after radiofrequency.
  Assessment of intensity of pain has been done in this order at:
  * Pre-selection visit: First algology assessment within a week (± 3 days) after the radiology consultation,
  * Inclusion visit: Second algology assessment (One week after the first algology assessment)
  * J-1: one day before radiofrequency
  * J+1: One day after radiofrequency
  * Discharge from hospital
  * 7 days after discharge from hospital
  * 1 month after radiofrequency
  * 2 months after radiofrequency
  * 3 months after radiofrequency
  Here, are presented only data collected one day before radiofrequency (J-1).
Time Frame: Algology assessment one day before radiofrequency (J-1)
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Patient Who Has Undergone Radiofrequency Ablation of Bone Metastases
Number analyzed (Participants) | 55
score on a scale
  Minimal pain | 2.0 (1.7)
  Average pain | 5.0 (1.7)
  Maximum pain | 7.0 (1.6)

6. Secondary Outcome: Intensity of Pain (Minimum, Average, Maximum)
Description: According to a discrete 11-points numerical scale which ranges from 0 (low pain) to 11 (intense pain), intensity of pain (Minimum, Average, Maximum) has been evaluated at different time point between pre-selection and up to 3 months after radiofrequency.
  Assessment of intensity of pain has been done in this order at:
  * Pre-selection visit: First algology assessment within a week (± 3 days) after the radiology consultation,
  * Inclusion visit: Second algology assessment (One week after the first algology assessment)
  * J-1: one day before radiofrequency
  * J+1: One day after radiofrequency
  * Discharge from hospital
  * 7 days after discharge from hospital
  * 1 month after radiofrequency
  * 2 months after radiofrequency
  * 3 months after radiofrequency
  Here, are presented only data collected one day after radiofrequency (J+1).
Time Frame: Algology assessment one day after radiofrequency: J+1
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Patient Who Has Undergone Radiofrequency Ablation of Bone Metastases
Number analyzed (Participants) | 55
score on a scale
  Minimal pain | 0.0 (1.6)
  Average pain | 2.0 (2.0)
  Maximum pain | 4.0 (2.7)

7. Secondary Outcome: Intensity of Pain (Minimum, Average, Maximum)
Description: According to a discrete 11-points numerical scale which ranges from 0 (low pain) to 11 (intense pain), intensity of pain (Minimum, Average, Maximum) has been evaluated at different time point between pre-selection and up to 3 months after radiofrequency.
  Assessment of intensity of pain has been done in this order at:
  * Pre-selection visit: First algology assessment within a week (± 3 days) after the radiology consultation,
  * Inclusion visit: Second algology assessment (One week after the first algology assessment)
  * J-1: one day before radiofrequency
  * J+1: One day after radiofrequency
  * Discharge from hospital
  * 7 days after discharge from hospital
  * 1 month after radiofrequency
  * 2 months after radiofrequency
  * 3 months after radiofrequency
  Here, are presented only data collected at the discharge from hospital visit.
Time Frame: Algology assessment at the discharge from hospital visit
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Patient Who Has Undergone Radiofrequency Ablation of Bone Metastases
Number analyzed (Participants) | 55
score on a scale
  Minimal pain | 0.0 (1.4)
  Average pain | 2.0 (1.8)
  Maximum pain | 3.0 (2.6)

8. Secondary Outcome: Intensity of Pain (Minimum, Average, Maximum)
Description: According to a discrete 11-points numerical scale which ranges from 0 (low pain) to 11 (intense pain), intensity of pain (Minimum, Average, Maximum) has been evaluated at different time point between pre-selection and up to 3 months after radiofrequency.
  Assessment of intensity of pain has been done in this order at:
  * Pre-selection visit: First algology assessment within a week (± 3 days) after the radiology consultation,
  * Inclusion visit: Second algology assessment (One week after the first algology assessment)
  * J-1: one day before radiofrequency
  * J+1: One day after radiofrequency
  * Discharge from hospital
  * 7 days after discharge from hospital
  * 1 month after radiofrequency
  * 2 months after radiofrequency
  * 3 months after radiofrequency
  Here, are presented only data collected 7 days after discharge from hospital.
Time Frame: Algology assessment 7 days after discharge from hospital
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Patient Who Has Undergone Radiofrequency Ablation of Bone Metastases
Number analyzed (Participants) | 55
score on a scale
  Minimal pain | 0.0 (2.0)
  Average pain | 2.0 (2.7)
  Maximum pain | 6.0 (3.1)

9. Secondary Outcome: Intensity of Pain (Minimum, Average, Maximum)
Description: According to a discrete 11-points numerical scale which ranges from 0 (low pain) to 11 (intense pain), intensity of pain (Minimum, Average, Maximum) has been evaluated at different time point between pre-selection and up to 3 months after radiofrequency.
  Assessment of intensity of pain has been done in this order at:
  * Pre-selection visit: First algology assessment within a week (± 3 days) after the radiology consultation,
  * Inclusion visit: Second algology assessment (One week after the first algology assessment)
  * J-1: one day before radiofrequency
  * J+1: One day after radiofrequency
  * Discharge from hospital
  * 7 days after discharge from hospital
  * 1 month after radiofrequency
  * 2 months after radiofrequency
  * 3 months after radiofrequency
  Here, are presented only data collected 1 month after radiofrequency.
Time Frame: Algology assessment 1 month after radiofrequency
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Patient Who Has Undergone Radiofrequency Ablation of Bone Metastases
Number analyzed (Participants) | 55
score on a scale
  Minimal pain | 0.0 (1.1)
  Average pain | 2.0 (2.0)
  Maximum pain | 3.0 (2.6)

10. Secondary Outcome: Intensity of Pain (Minimum, Average, Maximum)
Description: According to a discrete 11-points numerical scale which ranges from 0 (low pain) to 11 (intense pain), intensity of pain (Minimum, Average, Maximum) has been evaluated at different time point between pre-selection and up to 3 months after radiofrequency.
  Assessment of intensity of pain has been done in this order at:
  * Pre-selection visit: First algology assessment within a week (± 3 days) after the radiology consultation,
  * Inclusion visit: Second algology assessment (One week after the first algology assessment)
  * J-1: one day before radiofrequency
  * J+1: One day after radiofrequency
  * Discharge from hospital
  * 7 days after discharge from hospital
  * 1 month after radiofrequency
  * 2 months after radiofrequency
  * 3 months after radiofrequency
  Here, are presented only data collected 2 months after radiofrequency.
Time Frame: Algology assessment 2 months after radiofrequency
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Patient Who Has Undergone Radiofrequency Ablation of Bone Metastases
Number analyzed (Participants) | 55
score on a scale
  Minimal pain | 0.0 (1.1)
  Average pain | 2.0 (2.1)
  Maximum pain | 3.0 (2.7)

11. Secondary Outcome: Intensity of Pain (Minimum, Average, Maximum)
Description: According to a discrete 11-points numerical scale which ranges from 0 (low pain) to 11 (intense pain), intensity of pain (Minimum, Average, Maximum) has been evaluated at different time point between pre-selection and up to 3 months after radiofrequency.
  Assessment of intensity of pain has been done in this order at:
  * Pre-selection visit: First algology assessment within a week (± 3 days) after the radiology consultation,
  * Inclusion visit: Second algology assessment (One week after the first algology assessment)
  * J-1: one day before radiofrequency
  * J+1: One day after radiofrequency
  * Discharge from hospital
  * 7 days after discharge from hospital
  * 1 month after radiofrequency
  * 2 months after radiofrequency
  * 3 months after radiofrequency
  Here, are presented only data collected 3 months after radiofrequency.
Time Frame: Algology assessment 3 months after radiofrequency
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Patient Who Has Undergone Radiofrequency Ablation of Bone Metastases
Number analyzed (Participants) | 55
score on a scale
  Minimal pain | 0.0 (1.2)
  Average pain | 1.0 (2.3)
  Maximum pain | 2.5 (2.9)

12. Secondary Outcome: Oral Morphine Consumption or Oral Morphine Equivalent (Immediate and Sustained Release Forms) (mg) Per Day
Description: Patients were provided with a pain notebook. This notebook allowed the patient to describe the pain specific to the metastasis concerned.
  In particular, information about the dose of oral morphine consumption or oral morphine equivalent in mg per day.
  This pain notebook has been evaluated between the radiology consultation and three months after radiofrequency.
Time Frame: Preselection: First algology visit (within a week (± 3 days) after the radiology consultation)
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: mg morphine equivalents/day
Arm/Group | Patient Who Has Undergone Radiofrequency Ablation of Bone Metastases
Number analyzed (Participants) | 55
mg morphine equivalents/day | 60.0 (182.9)

13. Secondary Outcome: Oral Morphine Consumption or Oral Morphine Equivalent (Immediate and Sustained Release Forms) (mg) Per Day
Description: as for outcome 12
Time Frame: Inclusion: Second algology visit (One week after the first algology visit)
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: mg morphine equivalents/day
Arm/Group | Patient Who Has Undergone Radiofrequency Ablation of Bone Metastases
Number analyzed (Participants) | 55
mg morphine equivalents/day | 60.0 (182.9)

14. Secondary Outcome: Oral Morphine Consumption or Oral Morphine Equivalent (Immediate and Sustained Release Forms) (mg) Per Day
Description: as for outcome 12
Time Frame: J-1 (One day before radiofrequency)
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: mg morphine equivalents/day
Arm/Group | Patient Who Has Undergone Radiofrequency Ablation of Bone Metastases
Number analyzed (Participants) | 55
mg morphine equivalents/day | 60.0 (132.8)

15. Secondary Outcome: Oral Morphine Consumption or Oral Morphine Equivalent (Immediate and Sustained Release Forms) (mg) Per Day
Description: as for outcome 12
Time Frame: Discharge from hospital
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: mg morphine equivalents/day
Arm/Group | Patient Who Has Undergone Radiofrequency Ablation of Bone Metastases
Number analyzed (Participants) | 55
mg morphine equivalents/day | 60.0 (115.3)

16. Secondary Outcome: Oral Morphine Consumption or Oral Morphine Equivalent (Immediate and Sustained Release Forms) (mg) Per Day
Description: as for outcome 12
Time Frame: 7 days after discharge
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: mg morphine equivalents/day
Arm/Group | Patient Who Has Undergone Radiofrequency Ablation of Bone Metastases
Number analyzed (Participants) | 55
mg morphine equivalents/day | 60.0 (103.1)

17. Secondary Outcome: Oral Morphine Consumption or Oral Morphine Equivalent (Immediate and Sustained Release Forms) (mg) Per Day
Description: as for outcome 12
Time Frame: 1 month after radiofrequency
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: mg morphine equivalents/day
Arm/Group | Patient Who Has Undergone Radiofrequency Ablation of Bone Metastases
Number analyzed (Participants) | 55
mg morphine equivalents/day | 60.0 (148.0)

18. Secondary Outcome: Oral Morphine Consumption or Oral Morphine Equivalent (Immediate and Sustained Release Forms) (mg) Per Day
Description: as for outcome 12
Time Frame: 2 months after radiofrequency
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: mg morphine equivalents/day
Arm/Group | Patient Who Has Undergone Radiofrequency Ablation of Bone Metastases
Number analyzed (Participants) | 55
mg morphine equivalents/day | 60.0 (148.0)

19. Secondary Outcome: Oral Morphine Consumption or Oral Morphine Equivalent (Immediate and Sustained Release Forms) (mg) Per Day
Description: as for outcome 12
Time Frame: 3 months after radiofrequency
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: mg morphine equivalents/day
Arm/Group | Patient Who Has Undergone Radiofrequency Ablation of Bone Metastases
Number analyzed (Participants) | 55
mg morphine equivalents/day | 50.0 (169.5)

20. Secondary Outcome: Total Intravenous Morphine Dose (mg)
Description: Total intravenous dose of morphine 24 hours after the radiofrequency was assessed during the patient's hospital stay.
  As a reminder, the post-operative analgesic treatment included intravenous paracetamol (4 g / 24h) and patient-controlled analgesia (PCA).
Time Frame: 24 hours after radiofrequency
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: mg
Arm/Group | Patient Who Has Undergone Radiofrequency Ablation of Bone Metastases
Number analyzed (Participants) | 55
mg | 3.0 (72.4)

21. Secondary Outcome: Bolus Dose in mg Administered by Patient-controlled Analgesia (PCA)
Description: As a reminder, the post-operative analgesic treatment included intravenous paracetamol (4 g / 24h) and patient-controlled analgesia (PCA).
Time Frame: 24 hours after radiofrequency
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: mg
Arm/Group | Patient Who Has Undergone Radiofrequency Ablation of Bone Metastases
Number analyzed (Participants) | 55
mg | 1.0 (6.1)

22. Secondary Outcome: Standardised Quality of Life Scores (EORTC - QLQ-C30)
Description: Quality of life Questionnaire -Core 30 (QLQ-C30) developed in 1986 by the European Organization for Research and Treatment of Cancer (EORTC) assesses quality of life across 15 dimensions :
  5 functional dimensions : Physical functioning, Role functioning, Emotional, Cognitive functioning, Social functioning; 9 symptomatic dimensions: Fatigue, Nausea and vomiting, Pain, Dyspnea, Insomnia, Appetite loss, Diarrhoea, Financial difficulties;
  1 global health dimension: Global health status/QoL
  Each dimension is a standardised score ranges from 0 to 100. A low score corresponds to a low functional level, an absence of symptoms or a low level of QoL/ overall health and, conversely, so that a high score corresponds to a high functional level, a high presence of symptoms or a high level of QoL/overall health.
Time Frame: Inclusion
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Patient Who Has Undergone Radiofrequency Ablation of Bone Metastases
Number analyzed (Participants) | 55
score on a scale
  Physical functioning | 46.7 (23.7)
  Role functioning | 33.3 (32.9)
  Emotional functioning | 58.3 (24.2)
  Cognitive functioning | 66.7 (25.6)
  Social functioning | 33.3 (25.6)
  Global health status/QoL | 41.7 (17.1)
  Fatigue | 66.7 (23.1)
  Nausea and vomiting | 16.7 (26.5)
  Pain | 83.3 (24.4)
  Dyspnoea | 33.3 (30.6)
  Insomnia | 33.3 (31.5)
  Appetite loss | 0.0 (36.0)
  Constipation | 33.3 (33.1)
  Diarrhoea | 0.0 (16.3)
  Financial difficulties | 0.0 (26.3)

23. Secondary Outcome: Standardised Quality of Life Scores (EORTC - QLQ-C30)
Description: as for outcome 22
Time Frame: 2 months after radiofrequency
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Patient Who Has Undergone Radiofrequency Ablation of Bone Metastases
Number analyzed (Participants) | 55
score on a scale
  Physical functioning | 60.0 (23.9)
  Role functioning | 50.0 (29.9)
  Emotional functioning | 62.5 (20.8)
  Cognitive functioning | 50.0 (25.5)
  Social functioning | 50.0 (33.7)
  Global health status/QoL | 50.0 (19.0)
  Fatigue | 55.6 (25.7)
  Nausea and vomiting | 0.0 (21.3)
  Pain | 50.0 (28.2)
  Dyspnoea | 33.3 (33.2)
  Insomnia | 33.3 (35.0)
  Appetite loss | 33.3 (35.0)
  Constipation | 33.3 (37.4)
  Diarrhoea | 0.0 (23.8)
  Financial difficulties | 0.0 (16.9)

ADVERSE EVENTS:
Time Frame: All expected (SAE-E) and unexpected (SAE-U) serious adverse events, whether or not attributable to the research, that occur during the study or within 30 days afterwards. A serious adverse event report form (initial or follow-up) must be completed. According to the context Adverse Event (AE) not including serious has not been collected for this study.
Description: Adverse Event (AE) not including serious has not been collected for this study.
Arm/Group | Patient Who Has Undergone Radiofrequency Ablation of Bone Metastases
All-Cause Mortality (participants affected / at risk) | 10/71
Serious Adverse Events (participants affected / at risk) | 33/71
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patient Who Has Undergone Radiofrequency Ablation of Bone Metastases (N=71)
Febrile aplasia (Blood and lymphatic system disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 11 (11)
Alteration of the general condition (General disorders) | 10 (10)
Disease-related death (General disorders) | 3 (3)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fever (General disorders) | 1 (1) — Febrile syndrome (in the absence of neutropenia, where neutropenia is defined as absolute neutrophil count (ANC) <1.0 x 10e9/L)
Fracture (Injury, poisoning and procedural complications) | 6 (6)
Anemia (Blood and lymphatic system disorders) | 5 (9)
Jaundice (Hepatobiliary disorders) | 1 (1) — Compression of the bile ducts
Sciatalgy (Nervous system disorders) | 2 (3)
Immediate post-operative pain increase (Injury, poisoning and procedural complications) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1)
Dysuric syndrome (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes